CLINICAL TRIAL: NCT00968409
Title: Labeling of Receptor Ligands and Other Compounds With Halogen Radionuclides: Assessment of Progesterone Receptors in Breast Carcinoma by Positron Emission Tomography (PET) Using FFNP
Brief Title: Assessment of Progesterone Receptors in Breast Carcinoma by Positron Emission Tomography (PET) Using Fluoro Furanyl Norprogesterone (FFNP)
Acronym: FFNP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Principal Investigator, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FFNP 06-1034
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hormone Receptor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FFNP-PET/CT Imaging (Other): All subjects will receive an injection of F-18-FFNP followed by PET/CT imaging, laboratory testing and safety testing.
  Interventions: Radiation: PET; Other: Laboratory Testing; Other: Safety Testing; Drug: F18-FFNP

INTERVENTIONS:
Radiation: PET — PET imaging following injection of F18-FFNP to image hormone receptor status in patients with newly diagnosed breast cancer
Other: Laboratory Testing — Blood and urine samples for standard laboratory testing and radioactive counts will be obtained during the imaging sessions. Testing will include: urinalysis, complete blood count, comprehensive metabolic panel, and progesterone levels
Other: Safety Testing — ECG tracings and vital signs (blood pressure, heart rate, body temperature and respiration rate) are obtained at several time points before, during and after the imaging sessions.
Drug: F18-FFNP — injection of F18-FFNP

SUMMARY:
The purpose of this study is to see if Positron Emission Tomography (PET) imaging with a radioactive form of the hormone progesterone called FFNP will give the same results as hormone receptor testing already performed on tissue used to diagnose breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Biopsy-proven breast cancer
* Tumor estrogen-receptor and progesterone-receptor status already determined or scheduled to be determined at time of surgery without intervening therapy.
* Primary lesion size ≥ 1.5 cm as determined by imaging studies (ultrasonography, mammography, CT or MRI) or physical examination
* Able to give informed consent
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and / or documented hysterectomy), post menopausal (cessation of menses for more than 1 year), non lactating, or of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of FFNP) is negative.

Exclusion Criteria:

* No previous history of hormone therapy; NOTE - subjects who were treated with hormone therapy for reasons other than breast cancer or breast cancer prevention may be allowed to participate after review of history by the primary investigator
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of the other cancer present within the last 5 years
* Unable to tolerate 60-90 minutes of PET imaging per imaging session

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of FFNP-PET imaging compared to in-vivo receptor status | 4 years

SECONDARY OUTCOMES:
To assess the diagnostic quality of FFNP-PET images at the proposed 10.0 mCi dose | 4 years
To determine the relationship between tumor FFNP uptake and in vitro status of progesterone receptor | 4 years
To calculate human dosimetry and overall safety of FFNP-PET imaging | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University / Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Result] Dehdashti F, Laforest R, Gao F, Aft RL, Dence CS, Zhou D, Shoghi KI, Siegel BA, Katzenellenbogen JA, Welch MJ. Assessment of progesterone receptors in breast carcinoma by PET with 21-18F-fluoro-16alpha,17alpha-[(R)-(1'-alpha-furylmethylidene)dioxy]-19-norpregn-4-ene-3,20-dione. J Nucl Med. 2012 Mar;53(3):363-70. doi: 10.2967/jnumed.111.098319. Epub 2012 Feb 13. PMID 22331216